CLINICAL TRIAL: NCT06597734
Title: A Phase 2 Study Evaluating Olutasidenib in Combination With Hypomethylating Agents in Patients With IDH1-mutated Higher-risk Myelodysplastic Syndromes, Chronic Myelomonocytic Leukemia, or Advanced Myeloproliferative Neoplasm
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0515; NCI-2024-07758 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Chronic Myelomonocytic Leukemia; Advanced Myeloproliferative Neoplasms; IDH1-mutated Higher-Risk Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — olutasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olutasidenib+Azacitidine-IV or SubQ (Experimental): Participants will take capsules of olutasidenib 2 times each day while you are on study. Each dose should be taken about 12 hours apart at least 1 hour before or 2 hours after a meal. Azacitidine IV or Sub Q for 7 days every 28 days.
  Interventions: Drug: Olutasidenib

INTERVENTIONS:
Drug: Olutasidenib — Given by PO

SUMMARY:
To learn if olutasidenib, when combined with a drug called a hypomethylating agent (HMA) can help to control MDS, CMML, and/or MPN. The safety of the drug combination will also be studied.

DETAILED DESCRIPTION:
Primary Objectives To determine the overall response rate of olutasidenib in combination with investigator's choice of HMA in patients with IDH1-mutated higher-risk MDS/CMML or advanced MPN Secondary Objectives

The secondary objectives of this study are:

* To evaluate the rates of complete remission (CR) and median duration of CR
* To ascertain the safety and tolerability of olutasidenib with HMA in this participant population
* To determine survival including overall survival (OS), progression-free survival (PFS), and duration of response (DOR) To analyze reduction in IDH1 clone size Exploratory Objectives
* To examine overall response rate of patients previously exposed to venetoclax
* To investigate global gene expression profiles, DNA methylation profiles, and other potential prognostic markers to explore predictors of antitumor activity and/or resistance to treatment

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven higher-risk MDS/CMML or advanced MPN

   1. MDS participants must have International Prognostic Scoring System (IPSS) intermediate-2- or high-risk disease or Revised IPSS (IPSS-R) score >= 3.5 or Molecular IPSS (IPSS-M) moderate high-, high-, or very high-risk disease or bone marrow blast percentage.
   2. CMML patients must have CPSS-Mol int-1, int-2, or high-ris disease (Elena C et al, Blood 2016)
   3. Advanced MPN is defined as bone marrow blast percentage >=/=10%.
   4. Participants on the treatment-naive arm must not have received a prior HMA. Agents such as growth factors (e.g. erythropoietin stimulating agents, luspatercept, eltrombopag, granulocyte colony stimulating factors), cyclosporine, and/or hydroxyurea are allowed.
   5. Patients on the previously-treated arm must have received a prior HMA and/or ivosidenib. Prior stem cell transplantation in allowed>
2. Participants must have a documented IDH1 mutation
3. Patients with previously-treated MDS must be ineligible to receive treatment with ivosidenib or have progressed on treatment with ivosidenib.
4. Participants >=/= 18 years old
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 (Appendix A)
6. Acceptable liver function

   1. Bilirubin </= 2 times upper limit of normal (ULN) or <;/= 3 times ULN in participants with Gilbert Syndrome
   2. Aspartate transaminase (AST), alanine transaminase (ALT), and alkaline phosphatase </= 3 times ULN
7. Acceptable renal function calculated creatinine clearance >/= 50 mL/min (as assessed by Cockcroft-Gault, MDRD, or CKD-Epi validated measures)
8. Negative serum or urine pregnancy test if female of childbearing potential c. For fertile men and women, agreement to use highly effective contraceptive methods for the duration of study participation and 90 days after the last dose of study medication d. Agreement for male participants not to donate sperm and for female participants of childbearing potential not to donate ova during the study and for 90 days after the final dose of study drug
9. Ability and willingness to sign informed consent prior to beginning study and undergoing procedures

Exclusion Criteria:

1. Participants unable to swallow oral medications, or participants with gastrointestinal conditions (e.g., malabsorption, resection, etc.) deemed by the Investigator to jeopardize intestinal absorption
2. Participants with any concurrent uncontrolled clinically significant medical condition, including life-threatening severe infection or psychiatric illness, which could place the participant at unacceptable risk of study treatment
3. Patients must have discontinued prior chemotherapy at least 1 week prior to the start of study treatment. Patients with MPN must be off JAK inhibitors at the start of study treatment
4. Patients with active graft-versus-host-disease (GVHD) status post stem cell transplantation, including active chronic GVHD requiring topical therapy. Patients must have discontinued calcineurin inhibitors at least 4 weeks prior to the start of study treatment
5. Known active hepatitis B (HBV) or hepatitis C (HCV) or HIV infection
6. Pregnant or nursing women or women of childbearing potential not using highly effective contraception; male participants not using highly effective contraception
7. Participants with white blood cell count > 25 x109/L Note: hydroxyurea use is permitted to meet this criterion
8. Unwillingness or inability to comply with procedures either required in this protocol or considered standard of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Chien, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — https://www.mdanderson.org